CLINICAL TRIAL: NCT07019987
Title: Imaging the Respiratory Effects of Truncal Adiposity in Acute Hypoxemic Respiratory Failure
Brief Title: Adiposity Distribution in Acute Respiratory Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maurizio F. Cereda, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Maurizio F. Cereda, MD, Associate Professor of Anesthesia, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025P001410
Record Dates: First submitted 2025-05-20; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Acute Hypoxemic Respiratory Failure; Obesity
Keywords: acute hypoxemic respiratory failure; obesity; electrical impedance tomography; esophageal manometry; mechanical ventilation; prone positioning; positive end expiratory pressure
MeSH Terms: conditions — Respiratory Insufficiency; Obesity | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: In a prospective, single-center, physiological, crossover study, the investigators will recruit 80 mechanically ventilated adults with acute hypoxemic respiratory failure, across four standard body mass index categories (normal weight, overweight, class I obesity, class II/III obesity) and sex.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Ventilatory Assessment at Two PEEP Levels and Body Positions (Experimental): A total of 80 patients will undergo sequential assessments during mechanical ventilation at two levels of PEEP:
  1. Clinician-set PEEP (PEEP_CLIN)
  2. PEEP determined by EIT-guided titration (PEEP_TIT) These interventions will be applied first in the supine position, with each PEEP level maintained for approximately 30 minutes. Afterward, patients will be repositioned to the prone position, and the same assessments and EIT-guided PEEP titration will be repeated.
  Interventions: Other: PEEP Titration Using Electrical Impedance Tomography (EIT); Procedure: Body Positioning: Supine and Prone

INTERVENTIONS:
Other: PEEP Titration Using Electrical Impedance Tomography (EIT) — EIT will be used to guide individualized PEEP titration in mechanically ventilated patients with AHRF. Each subject will receive mechanical ventilation at two PEEP levels:
  PEEP_CLIN (set by the treating clinician)
  PEEP_TIT (identified using EIT to minimize alveolar collapse and overdistension)
  Both levels will be maintained for 30 minutes in each body position, with continuous physiologic data collected during each phase.
Procedure: Body Positioning: Supine and Prone — Each subject will be ventilated in both the supine and prone positions. Positioning will follow institutional protocols and be coordinated with clinical staff to ensure safety. After supine assessments are completed, the patient will be transitioned to prone, followed by a recruitment maneuver to standardize lung volume history. The PEEP titration protocol will then be repeated in the prone position.

SUMMARY:
Acute Hypoxemic Respiratory Failure (AHRF) is a condition in which injury to the lungs impairs the ability of the air sacs (alveoli) to ventilate and exchange oxygen. This impairment may be worsened in individuals with elevated body weight, particularly when fat tissue compresses the lungs and promotes alveolar collapse. The impact of body weight on lung function may be greater in individuals with upper-body fat distribution.

Two common interventions for AHRF-positive end-expiratory pressure (PEEP) and prone positioning-are used to improve lung ventilation. However, it is unclear whether these therapies are equally effective across different body weight categories and fat distributions.

This study will evaluate whether body weight and fat distribution affect patients' lung inflation responses to PEEP and prone positioning. Lung inflation will be assessed using electrical impedance tomography (EIT), a bedside imaging tool that maps lung ventilation, and esophageal manometry, which estimates lung compression through a thin catheter placed in the esophagus. Laboratory tests will also be used to measure markers of inflammation and AHRF severity and find correlations with fat distribution and responses to the tested treatments..

Patients with AHRF requiring mechanical ventilation will be enrolled across a range of body weights. Each participant will undergo combinations of two PEEP levels and two body positions (supine and prone) for 30 minutes each. At the end of the study procedures, clinical care will continue as determined by the treating team.

DETAILED DESCRIPTION:
This study investigates the relationship between body habitus and the physiological response to ventilatory interventions in patients with Acute Hypoxemic Respiratory Failure (AHRF). The primary objectives are to determine:

1. Whether excess body weight affects the regional lung inflation response to PEEP and prone positioning;
2. Whether body fat distribution (e.g., central vs. peripheral) is associated with lung recruitment;
3. Whether inflation responses correlate with laboratory markers of systemic inflammation and AHRF severity.

Adult patients with AHRF requiring invasive mechanical ventilation will be screened daily in the intensive care units at Massachusetts General Hospital. The study team will coordinate with clinical staff and patient surrogates to obtain informed consent. Enrollment is limited to the period required to perform study-specific procedures. No follow-up visits or post-discharge interventions are planned.

After consent, participants will be equipped with two adhesive EIT electrode belts, placed bilaterally on the thorax, to measure regional ventilation. A pressure and flow sensor will be placed in the breathing circuit at the proximal end of the endotracheal tube. An esophageal balloon catheter will be inserted nasally into the distal esophagus (approximately 35-40 cm) to measure intrathoracic pressure (ITP) via esophageal manometry, recorded through an auxiliary module on the EIT device.

Once all monitoring devices are in place, patients will be evaluated for adequate sedation and ventilator synchrony. Baseline data will be recorded during ventilation at the clinician-selected PEEP level (PEEP_CLIN), including EIT, airway pressure, flow, and ITP signals over 20 consecutive breaths.

Subsequently, a PEEP titration trial will be conducted to identify an individualized PEEP value (PEEP_TIT) that minimizes both alveolar collapse and overdistension, using EIT-based criteria. The patient will then be ventilated at PEEP_TIT for 30 minutes, after which all measurements will be repeated.

Following supine data collection, patients will be transitioned to the prone position using standard clinical protocols, with participation from ICU staff (physicians, nurses, and respiratory therapists) in accordance with institutional practice. Continuous monitoring (including pulse oximetry and arterial blood pressure) will be maintained throughout the repositioning.

After achieving the prone position, a recruitment maneuver will be performed to standardize lung volume history. The EIT belts will then be reconnected, and the patient will be allowed to stabilize for 30 minutes at PEEP_CLIN before measurements are repeated. A second PEEP titration trial will be performed to determine PEEP_TIT in the prone position, followed by another 30-minute stabilization period and repeat data acquisition.

Arterial blood samples (2 mL each) will be obtained at each PEEP level in both positions (four total, 8 mL cumulative) for gas exchange analysis. An additional 10 mL sample will be collected during supine ventilation at PEEP_CLIN for biomarker analysis. Biomarkers of inflammation (e.g., IL-6, TNF-α, C-reactive protein) and adipose tissue-related factors (e.g., adiponectin, leptin, resistin) will be measured.

After study procedures, participants will be returned to the supine position unless otherwise indicated by the clinical team. All subsequent clinical decisions regarding ventilator management or patient positioning will be made by the attending care team.

This study seeks to generate mechanistic insights into how excess body weight and fat distribution affect the physiologic response to standard ventilatory interventions in AHRF, with the goal of informing more individualized approaches to respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* AHRF with PaO2/FiO2 <= 300 mmHg) intubated for less than 72 hours
* Presence of an arterial line for blood gas measurement and blood pressure monitoring
* 18 years or older

Exclusion Criteria:

* Suspected pregnancy, pregnancy or less than six weeks postpartum
* Younger than 18 years or older than 80 years.
* Subject enrolled in another interventional research study
* Presence of pneumothorax
* Usage of any devices with electric current generation such as pacemaker or internal cardiac defibrillator
* Preexisting chronic lung disease or pulmonary hypertension
* Acute cardiac failure causing pulmonary edema
* Past medical history of lung malignancy or pneumonectomy, or lung transplant
* Hemodynamic instability, defined as:

  * Persistent systolic blood pressure <90 mmHg and/or >180 mmHg despite the use of vasopressor or vasodilators, or
  * Requiring an increment in inotropic-vasopressors over the past two hours just before enrollment: more than 15 mcg/min for norepinephrine and dopamine, more than 10 mcg/min in epinephrine; and more than 50 mcg/ min for phenylephrine.
* Contraindications to placement in the prone position: complex abdominal surgical dressing, recent sternotomy, unstable spine or pelvic fractures, intracranial hypertension, serious facial injury
* Extracorporeal life support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Driving pressure with PEEP titration and prone position | Day 1, after 30 minutes in each combination of PEEP and body position
  The primary outcome will be the difference in driving pressure (inspiratory plateau pressure minus total PEEP, in cmH2O) in response to PEEP titration strategies and to prone position. Changes in driving pressure will be correlated with body mass index, and with measurements of thoracic, and abdominal circumference.

SECONDARY OUTCOMES:
Regional ventilation | Day 1, after 30 minutes in each combination of PEEP and body position
  Changes in EIT-derived measurements of regional ventilation with PEEP titration and prone positioning. EIT regional ventilation is measured as percentage of total ventilation in each examined lung region.

OTHER OUTCOMES:
Age | Day 1
  Age will be measured in years.
Height | Day 1
  Body height will be measured in meters and will be aggregated with body weight to yield body mass index (BMI) in kg/m^2.
Weight | Day 1
  Body weight will be measured in kg and will be aggregated with height to yield body mass index (BMI) in kg/m^2
Thoracic circumference | Day 1
  Thoracic circumference will be measured in cm using a tape ruler placed at nipple level.
Abdominal circumference | Day 1
  Abdominal circumference will be measured in cm using a tape ruler at the level of the umbilicus.
Hip circumference | Day1
  Hip circumference will be measured in cm using a tape ruler placed around the widest portion of the hips.
Comorbidities | Day 1
  The medical record will be reviewed and the presence of the following coexisting conditions will be recorded:
  Hypertension Diabetes Heart failure Liver disease Cancer
APACHE II | First 24 hours since admission
  APACHE II is a severity score (Crit Care Med. 1985 Oct;13(10):818-29.) that will result from the aggregation of the following variables obtained from the medical record on the day of the study:
  age, temperature, mean arterial pressure, pH, heart rate, respiratory rate, plasma sodium, potassium, creatinine, presence of acute renal failure (yes/no), hematocrit, white blood cell count, Glasgow coma scale, and inspired fraction of oxygen (<50%, >=50%).
AHRF etiology | Day 1
  The etiology of AHRF will be recorded from the medical record as a binary variable (pulmonary vs. non pulmonary cause).
Partial Pressure of Oxygen (PaO2) | Day 1, arterial blood gas samples will be taken at 4 time points, after 30 minutes in each combination of PEEP and body position
  The PaO2 will be measured in mmHg in arterial blood samples.
Arterial Partial Pressure of Carbon Dioxide (PCO2) | Day 1, arterial blood gas samples will be taken at 4 time points, after 30 minutes in each combination of PEEP and body position
  The PaCO2 will be measured in mmHg in arterial blood samples.
pH | Day 1, arterial blood gas samples will be taken at 4 time points, after 30 minutes in each combination of PEEP and body position
  The pH will be measured in arterial blood samples.
Bicarbonate | Day 1, arterial blood gas samples will be taken at 4 time points, after 30 minutes in each combination of PEEP and body position
  The plasma bicarbonate will be measured in mEq/l with an arterial blood sample.
Plateau airway pressure | Day 1, after 30 minutes in each combination of PEEP and body position
  Plateau airway pressure will be measured in cmH2O during an inspiratory hold of the ventilator.
Respiratory Rate | Day 1, after 30 minutes in each combination of PEEP and body position
  Respiratory rate will be measured in breaths per minute during tidal ventilation.
Peak inspiratory pressure | Day 1, after 30 minutes in each combination of PEEP and body position
  Peak inspiratory pressure will be measured in cmH2O at the end of a tidal breath by the ventilator.
Total positive end expiratory pressure (PEEPt) | Day 1, after 30 minutes in each combination of PEEP and body position
  PEEPt will be measured in cmH2O during an expiratory hold of the ventilator
Mean Arterial Blood Pressure | Day 1, after 30 minutes in each combination of PEEP and body position
  Mean arterial blood pressure will be measured in mmHg through a preexisting arterial line and recorded by the clinical monitor.
Vasoactive medications (dopamine, dobutamine, epinephrine, levosimendan, milrinone, vasopressin, norepinephrine) | Day 1
  We will calculate the Vasoactive-inotropic score (VIS). The VIS compares different vasoactive-inotropic drugs and doses among the patients. VIS = dopamine dose (mg/kg/min)+ dobutamine [mg/kg/min) +100 x epinephrine dose (mg/ kg/min) +50 x levosimendan dose [mg/kg/min) + 10 x milrinone dose [mg/kg/min)+ 10,000 x vasopressin [units/kg/min) + 100x norepinephrine dose [mg/kg/min) using the maximum dosing rates of vasoactive and inotropic medications. Ref: Koponen et al. British Journal of Anaesthesia, 122 (4): 428e436 (2019). This exploratory outcome plans to combine driving pressure and electrical impedance tomography with other markers (demographical, body metrics, clinical, biochemical, and inflammatory) to identify responses to PEEP and prone positioning.
Life Sustaining Therapies | Day 1
  The presence of the following life sustaining therapy on the day of the study (in addition to mechanical ventilation and vasoactive medications) will be recorded as binary variables (yes/no) from the medical record:
  antibiotics, renal replacement therapy, and artificial nutrition.
Interleukin 6 (IL-6) | Day 1, once
  IL-6 (ng/mL) is an inflammatory biomarker that will be measured in blood samples that will be collected on the day of the study.
C-reactive protein (CRP) | Day 1, once
  CRP (mg/L) is an inflammatory biomarker that will be measured on a blood sample obtained on the day of the study.
Adiponectin | Day 1, once
  Adiponectin (micrograms/mL) is a marker of adipose cell metabolic activity that will be measured in a blood sample obtained on the day of the study.
Leptin | Day 1, once
  Leptin (ng/mL) is a parker of adipose metabolic and proinflammatory activity that will be measured on a blood sample on the day of the study
Resistin | Day 1, once
  Resistin (ng/mL) is a marker of inflammatory activity secreted by adipose tissue, it will be measured in blood samples obtained on the day of the study.
tumor necrosis factor-alpha (TNF-alpha) | Day 1, once
  TNF alpha (picograms/mL) is an inflammatory biomarker that will be meaured in a blood sample obtained the day of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao D, Low S, Di Fenza R, Shenoy ES, Ananian L, Prout LA, La Vita CJ, Berra L. Prone Positioning of Intubated Patients with an Elevated Body-Mass Index. N Engl J Med. 2022 Apr 7;386(14):e34. doi: 10.1056/NEJMvcm2108494. No abstract available. PMID 35388669
- [Background] Kompaniyets L, Goodman AB, Belay B, Freedman DS, Sucosky MS, Lange SJ, Gundlapalli AV, Boehmer TK, Blanck HM. Body Mass Index and Risk for COVID-19-Related Hospitalization, Intensive Care Unit Admission, Invasive Mechanical Ventilation, and Death - United States, March-December 2020. MMWR Morb Mortal Wkly Rep. 2021 Mar 12;70(10):355-361. doi: 10.15585/mmwr.mm7010e4. PMID 33705371
- [Background] Behazin N, Jones SB, Cohen RI, Loring SH. Respiratory restriction and elevated pleural and esophageal pressures in morbid obesity. J Appl Physiol (1985). 2010 Jan;108(1):212-8. doi: 10.1152/japplphysiol.91356.2008. Epub 2009 Nov 12. PMID 19910329
- [Background] De Santis Santiago R, Teggia Droghi M, Fumagalli J, Marrazzo F, Florio G, Grassi LG, Gomes S, Morais CCA, Ramos OPS, Bottiroli M, Pinciroli R, Imber DA, Bagchi A, Shelton K, Sonny A, Bittner EA, Amato MBP, Kacmarek RM, Berra L; Lung Rescue Team Investigators. High Pleural Pressure Prevents Alveolar Overdistension and Hemodynamic Collapse in Acute Respiratory Distress Syndrome with Class III Obesity. A Clinical Trial. Am J Respir Crit Care Med. 2021 Mar 1;203(5):575-584. doi: 10.1164/rccm.201909-1687OC. PMID 32876469
- [Background] Florio G, De Santis Santiago RR, Fumagalli J, Imber DA, Marrazzo F, Sonny A, Bagchi A, Fitch AK, Anekwe CV, Amato MBP, Arora P, Kacmarek RM, Berra L. Pleural Pressure Targeted Positive Airway Pressure Improves Cardiopulmonary Function in Spontaneously Breathing Patients With Obesity. Chest. 2021 Jun;159(6):2373-2383. doi: 10.1016/j.chest.2021.01.055. Epub 2021 May 8. PMID 34099131
- [Background] Spina S, Mantz L, Xin Y, Moscho DC, Ribeiro De Santis Santiago R, Grassi L, Nova A, Gerard SE, Bittner EA, Fintelmann FJ, Berra L, Cereda M. The pleural gradient does not reflect the superimposed pressure in patients with class III obesity. Crit Care. 2024 Sep 16;28(1):306. doi: 10.1186/s13054-024-05097-6. PMID 39285477